CLINICAL TRIAL: NCT00425555
Title: A Phase II Study of Oral LBH589 in Adult Patients With Refractory Cutaneous T-Cell Lymphoma
Brief Title: Study of Oral LBH589 in Adult Patients With Refractory Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2201; 2006-000880-27 (EudraCT Number)
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cutaneous T-Cell Lymphoma
Keywords: Cutaneous T-Cell Lymphoma, adults; Mycosis Fungoides; Sézary Syndrome; CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Panobinostat

ARMS (2):
- Previously treated with oral bexarotene (Experimental): Participants received Panobinostat 20 milligrams per day (mg/day) capsule orally, once a day (OD) on 3 days per week. (Monday, Wednesday and Friday or alternative Day 1, 3 and 5).
  Interventions: Drug: Panobinostat
- No prior oral bexarotene treatment (Experimental): Participants received Panobinostat 20 milligrams per day (mg/day) capsule orally, once a day (OD) on 3 days per week. (Monday, Wednesday and Friday or alternative Day 1, 3 and 5).
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat
  Other Names: LBH589

SUMMARY:
This study will evaluate the safety and efficacy of LBH489B in adult patients with refractory Cutaneous T-Cell Lymphoma.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent obtained prior to any screening procedures
2. Age ≥ 18 years old
3. Patients with biopsy-confirmed stages IB-IVA mycosis fungoides or Sézary syndrome. Patients with SS who have bone marrow involvement are also eligible.
4. Patients must have received at least two prior treatment regimens at least one of which was a systemic therapy regimen. Systemic regimens include oral bexarotene, PUVA, photophoresis, oral corticosteroids, total skin electron bean therapy, chemotherapy such as methotrexate, and interferon. Topical steroids alone are not considered as a treatment regimen.
5. Patients must have had disease progression on or following their most recent treatment regimen or an inadequate response to their most recent treatment regimen.
6. Patients will be accrued to one of two groups: Patients previously treated with oral bexarotene and patients who have not had prior oral bexarotene treatment.

Exclusion criteria:

1. Prior treatment with an HDAC inhibitor.
2. Patients with visceral disease including CNS involvement (i.e. stage IVB CTCL). Note; Patients with SS who have bone marrow involvement are eligible.
3. Impaired cardiac function
4. Concomitant use of drugs with a risk of causing torsades de pointes
5. Patients who have received chemotherapy or any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
6. Less than 3 months since prior electron beam therapy
7. Female patients who are pregnant or breast feeding, or patients of reproductive potential not using an effective method of birth control, and male patients whose sexual partners are women of childbearing potential not using effective birth control
8. Uncontrolled hypertension
9. Concomitant use of any anti-cancer therapy or radiation therapy. Low potency topical steroid use is permitted. Topical bexarotene use is prohibited during the trial
10. Concomitant use of CYP3A4/5 inhibitors.
11. Patients with unresolved diarrhea > CTCAE grade 1
12. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
13. Other concurrent severe and/or uncontrolled medical conditions
14. Patients who would need to receive valproic acid for any reason during the study or ≤ 5 days prior to starting study drug.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2007-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (41):
- United States (16):
  - University of Alabama at Birmingham/ Kirklin Clinic Kirklin Clinic, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of California at Los Angeles Dept. of Hematology-Oncology, Los Angeles, California
  - Florida Academic Dermatology Center, Miami, Florida
  - Emory University School of Medicine/Winship Cancer Institute Dept. of Hematology (2), Atlanta, Georgia
  - Georgia Health Sciences University Dept.ofMedicalCollegeOfGeorgia, Augusta, Georgia
  - NorthwesternUniv.Med.School/Robert H. Lurie Comp.Cancer Ctr Dept. of NorthwesterUMed, Chicago, Illinois
  - Indiana University Dept. of IU Cancer Center, Indianapolis, Indiana
  - Boston Medical Center StudyCoordinator:CLBH589B2201, Boston, Massachusetts
  - Dana Farber Cancer Institute Deptof DanaFarberCancerInst(3), Boston, Massachusetts
  - University of Michigan Health System Michigan HouseClinTrialsOffice, Ann Arbor, Michigan
  - Wake Forest University Baptist Medical Center OutpatientCmprehensivCancerCtr, Winston-Salem, North Carolina
  - University Dermatology Consultants, Cincinnati, Ohio
  - Oregon Health & Science University Dept. of OHSU Cancer Institute, Portland, Oregon
  - University of Pittsburgh Medical Center Department of Dermatology, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center/University of Texas StudyCoordinator:CLBH589B2201, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (2):
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (3):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Yvoir
- Canada (2):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Helsinki, Finland
- France (3):
  - Novartis Investigative Site, Lyon, Cedex 02
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Paris
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Budapest, Hungary
- Italy (5):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland

REFERENCES:
- [Result] Duvic M, Dummer R, Becker JC, Poulalhon N, Ortiz Romero P, Grazia Bernengo M, Lebbe C, Assaf C, Squier M, Williams D, Marshood M, Tai F, Prince HM. Panobinostat activity in both bexarotene-exposed and -naive patients with refractory cutaneous T-cell lymphoma: results of a phase II trial. Eur J Cancer. 2013 Jan;49(2):386-94. doi: 10.1016/j.ejca.2012.08.017. Epub 2012 Sep 13. PMID 22981498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 41 centers in 12 countries.
Pre-assignment Details: A total 139 Participants were enrolled in the Study. No Patients completed treatment. All patients discontinued the treatment on this study and 136 patients discontinued the study (97.8%). The remaining three patients discontinued the study treatment were immediately transferred to another program.
Groups:
- Bexarotene Exposed; Bexarotene Naive: Participants received Panobinostat 20 milligrams per day (mg/day) capsule orally, once a day (OD) on 3 days per week. (Monday, Wednesday and Friday or alternative Day 1, 3 and 5). The treatment duration was not fixed. Participants continued treatment until disease progression or unacceptable toxicity occurred.
Period: Overall Study
Arm/Group | Bexarotene Exposed | Bexarotene Naive
Started | 79 | 60
Completed | 0 | 0
Not Completed | 79 | 60
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Administrative problems | 3 | 0
Not completed — Death | 1 | 2
Not completed — New cancer therapy | 2 | 1
Not completed — Disease progression | 36 | 33
Not completed — Adverse Event | 25 | 15
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed in Full analyses set (FAS) population was defined according to the intention-to-treat principle. This population will include all participants enrolled into the study.
Groups:
- Bexarotene Exposed; Bexarotene Naive: Participants received Panobinostat 20 mg/day capsule orally, OD on 3 days per week. (Monday, Wednesday and Friday or alternative Day 1, 3 and 5). The treatment duration was not fixed. Participants continued treatment until disease progression or unacceptable toxicity occurred.
- Total: Total of all reporting groups
Arm/Group | Bexarotene Exposed | Bexarotene Naive | Total
Number analyzed (Participants) | 79 | 60 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (14.70) | 62.1 (11.51) | 59.7 (13.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 19 | 51
  Male | 47 | 41 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 68 | 54 | 122
  Black | 3 | 3 | 6
  Asian | 3 | 1 | 4
  Other | 5 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Participants Using the Modified Severity-Weighted Assessment Tool (mSWAT)
Description: Skin response was primarily classified based on an assessment using mSWAT, provided there was documented evidence of stable disease or better in lymph node/viscera.The mSWAT is a tool specifically developed to evaluate the extent of skin disease in CTCL (Olsen et al 2007).
  Responses in the skin based on SWAT are defined as:
  * Complete Response (CR): no evidence of skin disease
  * Partial Response (PR): ≥ 50% decrease of the modified SWAT score compared with baseline
  * Stable Disease (SD): Neither CR, PR, or PD as compared with baseline, i.e. change from baseline is less than a 50% decrease but also less than a 25 % increase in the modified SWAT score
  * Progressive Disease (PD): ≥ 25% increase in the modified SWAT score compared with baseline.
Time Frame: Baseline up to 6 Months of Follow up
Population: The analysis was performed in Full Analysis Set (FAS) population was defined according to the intention-to-treat principle. This population will include all participants enrolled into the study.
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- All Participants: Participants received Panobinostat 20 mg/day capsule orally, OD on 3 days per week. (Monday, Wednesday and Friday or alternative Day 1, 3 and 5). The treatment duration was not fixed. Participants continued treatment until disease progression or unacceptable toxicity occurred.
Arm/Group | Bexarotene Exposed | Bexarotene Naive | All Participants
Number analyzed (Participants) | 79 | 60 | 139
percentage | 16.7 [8.1 to 25.0] | 20.3 [10.8 to 32.3] | 18.5 [11.4 to 24.6]

2. Secondary Outcome: The Overall Response Rate Using mSWAT Skin Score
Description: Estimate of the response rate of participants with resistant cutaneous T-cell lymphoma (CTCL) treated with Panobinostat using the mSWAT skin scores and 95% CI will be analyzed.
Time Frame: Baseline up to Cycle 12, an average of 12 months
Population: The analysis was performed in FAS population was defined according to the intention-to-treat principle. This population will include all participants enrolled into the study.
Measure: Count of Participants; unit: Participants
Groups:
- Bexarotene Exposed: Participants received Panobinostat 20 mg/day capsule orally, OD on 3 days per week. (Monday, Wednesday and Friday or alternative Day 1, 3 and 5). The treatment duration was not fixed.Participants continued treatment until disease progression or unacceptable toxicity occurred.
Arm/Group | Bexarotene Exposed | Bexarotene Naive | All Participants
Number analyzed (Participants) | 79 | 60 | 139
Participants
  mSWAT skin response (CR/PR)flare considered as disease progression ( f.i.p ) - Number of responders | 12 | 14 | 26
  Physician's Global Assessment- Responder (CR/PR) | 15 | 18 | 33

3. Secondary Outcome: Time to Response for Responders
Description: Time to response were summarized. A Kaplan-Meier analysis of time to progression was performed, including estimation and 95% confidence interval of the median time to progression and progression-free survival.
Time Frame: Baseline up to Cycle 12, an average of 12 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bexarotene Exposed | Bexarotene Naive | All Participants
Number analyzed (Participants) | 79 | 60 | 139
Days | 69.5 [29.0 to 141.0] | 85.5 [29.0 to 115.0] | 82.0 [30.0 to 113.0]

4. Secondary Outcome: Duration of Response (DOS)
Description: Duration of response and time to response were summarized. A Kaplan-Meier analysis of time to progression was performed, including estimation and 95% confidence interval of the median time to progression and progression-free survival.
Time Frame: Baseline up to Cycle 12, an average of 12 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Bexarotene Exposed | Bexarotene Naive | All Participants
Number analyzed (Participants) | 79 | 60 | 139
Days | 170.0 [86.0 to 294.0] | NA [84.0 to NA] — There were an insufficient number of participants with events and therefore the Median and Upper limit of the 95% CI for the duration of response could not be calculated. | 280.0 [115.0 to 311.0]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from first dose of study treatment to progression or death due to any cause, based on modified European Society for Bone and Marrow Transplantation (EBMT) criteria per Investigator's assessment
Time Frame: Baseline up to Cycle 12, an average of 12 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bexarotene Exposed | Bexarotene Naive | All Participants
Number analyzed (Participants) | 79 | 60 | 139
months | 127.0 [87.0 to 197.0] | 113.0 [85.0 to 142.0] | 114.0 [87.0 to 143.0]

6. Secondary Outcome: Skindex-29 Measurements of Average Sub-scores for Emotions From Baseline up to Cycle 12
Description: Skin index measurement (Skindex-29) was a self-administered 29-item dermatology patient-reported outcome measure that explores the domains of Functioning, Emotions and Symptoms. Data from the Skindex-29 came from the "Dermatology Survey" page. Scoring of the Skindex-29 was performed as per the developers' scoring algorithms. The score for each dimension was found by adding responses of 1 to 5 for each question, with higher scores indicating worse quality of life. The Skindex-29 yields three scale scores that assess emotions scores range from 29 to 116, with higher scores indicating worse health-related quality of life. Average sub-scores for emotions, physical symptoms, and functioning was displayed.
Time Frame: Baseline up to Cycle 12, an average of 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bexarotene Exposed | Bexarotene Naive
Number analyzed (Participants) | 79 | 60
score on a scale
  Baseline: number analyzed (Participants) | 79 | 57
  Baseline | 52.2 (22.66) | 50.6 (22.26)
  Cycle 2: number analyzed (Participants) | 71 | 53
  Cycle 2 | 48.6 (23.79) | 46.6 (24.18)
  Cycle 3: number analyzed (Participants) | 57 | 40
  Cycle 3 | 45.9 (21.53) | 44.1 (24.37)
  Cycle 4: number analyzed (Participants) | 40 | 29
  Cycle 4 | 40.8 (23.87) | 34.7 (21.59)
  Cycle 5: number analyzed (Participants) | 30 | 26
  Cycle 5 | 35.8 (22.19) | 34.4 (20.53)
  Cycle 6: number analyzed (Participants) | 25 | 24
  Cycle 6 | 34.5 (22.72) | 35.4 (20.74)
  Cycle 7: number analyzed (Participants) | 22 | 20
  Cycle 7 | 39.3 (24.98) | 36.8 (22.61)
  Cycle 8: number analyzed (Participants) | 17 | 17
  Cycle 8 | 39.4 (20.03) | 35.8 (22.39)
  Cycle 9: number analyzed (Participants) | 20 | 17
  Cycle 9 | 44.6 (23.09) | 32.8 (18.36)
  Cycle 10: number analyzed (Participants) | 18 | 13
  Cycle 10 | 43.6 (20.48) | 43.5 (24.10)
  Cycle 11: number analyzed (Participants) | 14 | 10
  Cycle 11 | 48.3 (20.92) | 43.5 (22.86)
  Cycle 12: number analyzed (Participants) | 11 | 8
  Cycle 12 | 42.0 (16.80) | 43.1 (21.29)

7. Secondary Outcome: Skindex-29 Measurements of Average Sub-scores for Functioning From Baseline up to Cycle 12
Description: Skindex-29 was a self-administered 29-item dermatology patient-reported outcome measure that explores the domains of Functioning, Emotions and Symptoms. Data from the Skindex-29 came from the "Dermatology Survey" page. Scoring of the Skindex-29 was performed as per the developers' scoring algorithms. The score for each dimension was found by adding responses of 1 to 5 for each question, with higher scores indicating worse quality of life. The Skindex-29 yields three scale scores that assess functioning scores range from 29 to 116, with higher scores indicating worse health-related quality of life. Average sub-scores for emotions, physical symptoms, and functioning was displayed.
Time Frame: Baseline up to Cycle 12, an average of 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bexarotene Exposed | Bexarotene Naive
Number analyzed (Participants) | 79 | 60
score on a scale
  Baseline: number analyzed (Participants) | 79 | 57
  Baseline | 46.7 (24.44) | 44.7 (25.33)
  Cycle 2: number analyzed (Participants) | 71 | 53
  Cycle 2 | 43.5 (26.27) | 43.3 (24.53)
  Cycle 3: number analyzed (Participants) | 57 | 40
  Cycle 3 | 42.6 (25.58) | 39.2 (26.38)
  Cycle 4: number analyzed (Participants) | 40 | 29
  Cycle 4 | 38.8 (25.91) | 30.7 (22.91)
  Cycle 5: number analyzed (Participants) | 30 | 26
  Cycle 5 | 32.8 (23.35) | 31.4 (21.38)
  Cycle 6: number analyzed (Participants) | 25 | 24
  Cycle 6 | 33.0 (27.79) | 29.5 (21.25)
  Cycle 7: number analyzed (Participants) | 22 | 20
  Cycle 7 | 33.1 (26.04) | 28.3 (22.98)
  Cycle 8: number analyzed (Participants) | 17 | 17
  Cycle 8 | 34.4 (22.73) | 30.5 (25.16)
  Cycle 9: number analyzed (Participants) | 19 | 17
  Cycle 9 | 37.2 (25.28) | 28.7 (19.54)
  Cycle 10: number analyzed (Participants) | 17 | 13
  Cycle 10 | 35.2 (25.21) | 41.5 (27.22)
  Cycle 11: number analyzed (Participants) | 14 | 10
  Cycle 11 | 40.0 (24.47) | 38.1 (25.46)
  Cycle 12: number analyzed (Participants) | 10 | 8
  Cycle 12 | 26.3 (12.79) | 36.2 (20.95)

8. Secondary Outcome: Skindex-29 Measurements of Average Sub-scores for Physical Symptoms From Baseline up to Cycle 12
Description: Skindex-29 was a self-administered 29-item dermatology patient-reported outcome measure that explores the domains of Functioning, Emotions and Symptoms. Data from the Skindex-29 came from the "Dermatology Survey" page. Scoring of the Skindex-29 was performed as per the developers' scoring algorithms. The score for each dimension was found by adding responses of 1 to 5 for each question, with higher scores indicating worse quality of life. The Skindex-29 yields three scale scores that assess physical symptoms scores range from 29 to 116, with higher scores indicating worse health-related quality of life. Average sub-scores for emotions, physical symptoms, and functioning was displayed.
Time Frame: Baseline up to Cycle 12, an average of 12 months
Population: The analysis was performed in FAS population was defined according to the intention-to-treat principle. This population included all participants enrolled into the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bexarotene Exposed | Bexarotene Naive
Number analyzed (Participants) | 79 | 60
score on a scale
  Baseline: number analyzed (Participants) | 78 | 57
  Baseline | 60.1 (19.03) | 55.3 (20.35)
  Cycle 2: number analyzed (Participants) | 70 | 53
  Cycle 2 | 51.4 (23.10) | 47.7 (20.28)
  Cycle 3: number analyzed (Participants) | 56 | 40
  Cycle 3 | 51.1 (21.92) | 42.9 (21.72)
  Cycle 4: number analyzed (Participants) | 40 | 29
  Cycle 4 | 47.3 (22.16) | 35.2 (16.66)
  Cycle 5: number analyzed (Participants) | 31 | 26
  Cycle 5 | 43.2 (23.96) | 35.6 (18.81)
  Cycle 6: number analyzed (Participants) | 26 | 24
  Cycle 6 | 43.5 (24.72) | 36.2 (19.02)
  Cycle 7: number analyzed (Participants) | 23 | 20
  Cycle 7 | 45.5 (23.67) | 37.7 (18.66)
  Cycle 8: number analyzed (Participants) | 18 | 17
  Cycle 8 | 42.7 (21.45) | 36.5 (19.29)
  Cycle 9: number analyzed (Participants) | 20 | 17
  Cycle 9 | 47.1 (23.42) | 35.9 (15.79)
  Cycle 10: number analyzed (Participants) | 18 | 13
  Cycle 10 | 46.8 (23.11) | 47.0 (21.17)
  Cycle 11: number analyzed (Participants) | 14 | 10
  Cycle 11 | 46.7 (22.04) | 48.3 (19.44)
  Cycle 12: number analyzed (Participants) | 11 | 8
  Cycle 12 | 37.7 (15.52) | 45.1 (21.93)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Panobinostat
Description: Cmax is defined as the maximum observed drug concentration observed in plasma over all PK sample concentrations. It will be obtained from the Cmax parameter calculated by WinNonlin®. If there is no measurable concentration in the subject's PK profile, then Cmax will be missing for that subject. Cmax will be reported in units of ng/mL.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: The analysis was performed in PK population, defined as all participants who provide at least one post-dose PK plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | All Participants
Number analyzed (Participants) | 139
ng/mL
  Day 1: number analyzed (Participants) | 109
  Day 1 | 11.379 (6.6608)
  Day 8: number analyzed (Participants) | 60
  Day 8 | 13.490 (6.4529)

10. Secondary Outcome: Time to Peak Concentration (Tmax) of Panobinostat
Description: Tmax is defined as the time at which the Cmax occurs. It will be obtained from the Tmax parameter calculated by WinNonlin®. If there is no measurable Cmax in the subject's PK profile, then Tmax will be missing for that subject. Tmax will be reported in units of h.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: The analysis was performed in PAS population, defined as all participants who provide at least one post-dose PK plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Median (Full Range); unit: h (hours)
Arm/Group | All Participants
Number analyzed (Participants) | 139
h (hours)
  Day 1: number analyzed (Participants) | 109
  Day 1 | 1.5 [0.00 to 4.00]
  Day 8: number analyzed (Participants) | 60
  Day 8 | 1.5 [0.25 to 3.50]

11. Secondary Outcome: Area Under the Plasma Concentration AUC0-24, AUC0-48 and AUC 0-infinity of Panobinostat
Description: AUC is defined as the area under concentration-time curve as a measure of drug exposure. The area under the plasma concentration-time curve from time zero to 24 hours. The area under the plasma concentration-time curve from time zero to 48 hours. AUC (0-inf) is defined as the area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | All Participants
Number analyzed (Participants) | 139
ng*hr/ml
  Day 1 - AUC0-24: number analyzed (Participants) | 109
  Day 1 - AUC0-24 | 110.138 (58.0235)
  Day 8 - AUC0-24: number analyzed (Participants) | 60
  Day 8 - AUC0-24 | 134.033 (61.5203)
  Day 1 - AUC0-48: number analyzed (Participants) | 107
  Day 1 - AUC0-48 | 132.019 (69.3453)
  Day 8 - AUC0-48: number analyzed (Participants) | 52
  Day 8 - AUC0-48 | 159.750 (64.2278)
  Day 1- AUC (0-inf): number analyzed (Participants) | 93
  Day 1- AUC (0-inf) | 134.828 (64.9389)
  Day 8 - AUC (0-inf): number analyzed (Participants) | 52
  Day 8 - AUC (0-inf) | 162.673 (65.0664)

12. Secondary Outcome: Time of Clast (Tlast) of Panobinostat
Description: Time of Clast (Tlast) will be obtained from the Tlast parameter calculated by WinNonlin®. If there is no measurable concentration in the subject's PK profile, then Tlast will be missing for that participants. Tlast will be reported in units of h.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | All Participants
Number analyzed (Participants) | 139
Hours
  Day 1: number analyzed (Participants) | 109
  Day 1 | 47.9 [23.40 to 49.50]
  Day 8: number analyzed (Participants) | 60
  Day 8 | NA [16.80 to 47.00] — below the level of detection

13. Secondary Outcome: Last Observed Plasma Concentration (Clast) of Panobinostat
Description: Clast is defined as the Last observed (quantifiable) plasma concentration (Clast), in units of ng/mL. Blood samples were collected to assess Clast.
Time Frame: Pre-dose, 0.25, 1-2, and 3-4 hours post dose on Day 1 and Day 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | All Participants
Number analyzed (Participants) | 139
ng/mL
  Day 1: number analyzed (Participants) | 109
  Day 1 | 0.632 (0.9737)
  Day 8: number analyzed (Participants) | 60
  Day 8 | 1.524 (0.9076)

ADVERSE EVENTS:
Time Frame: From Start of the Study up to 7 years approximately
Description: The analysis was performed on Safety analysis population (SAP) consisted of all participants who received at least one dose of study drug and had at least one valid post-baseline assessment.
Groups:
- Bexarotene Exposed; Bexarotene Naive: Participants received Panobinostat 20 mg/day capsule orally, OD on 3 days per week. (Monday, Wednesday and Friday or alternative Day 1, 3 and 5). Participants continued treatment until disease progression or unacceptable toxicity occurred.
Arm/Group | Bexarotene Exposed | Bexarotene Naive
All-Cause Mortality (participants affected / at risk) | 3/79 | 3/60
Serious Adverse Events (participants affected / at risk) | 33/79 | 23/60
Other Adverse Events (participants affected / at risk) | 77/79 | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene Exposed (N=79) | Bexarotene Naive (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 3 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 0
Hypothermia (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
Sudden cardiac death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Rotavirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 2
Skin bacterial infection (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Superinfection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bexarotene Exposed (N=79) | Bexarotene Naive (N=60)
Anaemia (Blood and lymphatic system disorders) | 17 | 6
Leukopenia (Blood and lymphatic system disorders) | 9 | 4
Neutropenia (Blood and lymphatic system disorders) | 14 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 40 | 23
Vertigo (Ear and labyrinth disorders) | 4 | 0
Hypothyroidism (Endocrine disorders) | 9 | 5
Conjunctivitis (Eye disorders) | 2 | 4
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 5
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3
Constipation (Gastrointestinal disorders) | 8 | 11
Diarrhoea (Gastrointestinal disorders) | 45 | 38
Dry mouth (Gastrointestinal disorders) | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 32 | 22
Vomiting (Gastrointestinal disorders) | 10 | 7
Asthenia (General disorders) | 22 | 10
Chills (General disorders) | 4 | 8
Fatigue (General disorders) | 26 | 29
Malaise (General disorders) | 4 | 5
Oedema peripheral (General disorders) | 10 | 12
Pyrexia (General disorders) | 12 | 8
Bronchitis (Infections and infestations) | 4 | 3
Cellulitis (Infections and infestations) | 0 | 4
Influenza (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 8 | 6
Skin infection (Infections and infestations) | 4 | 4
Urinary tract infection (Infections and infestations) | 7 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 4
Blood creatinine increased (Investigations) | 15 | 8
Blood triglycerides increased (Investigations) | 6 | 4
Blood urea increased (Investigations) | 6 | 1
Electrocardiogram QT prolonged (Investigations) | 5 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 4
Haemoglobin decreased (Investigations) | 5 | 3
Platelet count decreased (Investigations) | 4 | 4
Weight decreased (Investigations) | 10 | 6
Decreased appetite (Metabolism and nutrition disorders) | 19 | 17
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 11 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 14 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3
Dizziness (Nervous system disorders) | 10 | 6
Dysgeusia (Nervous system disorders) | 13 | 12
Headache (Nervous system disorders) | 16 | 12
Paraesthesia (Nervous system disorders) | 4 | 2
Somnolence (Nervous system disorders) | 2 | 4
Syncope (Nervous system disorders) | 4 | 2
Depression (Psychiatric disorders) | 4 | 7
Insomnia (Psychiatric disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 4
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 16
Rash (Skin and subcutaneous tissue disorders) | 4 | 4
Skin exfoliation (Skin and subcutaneous tissue disorders) | 7 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 6 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 4
Hypertension (Vascular disorders) | 11 | 4
Hypotension (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes